CLINICAL TRIAL: NCT06654128
Title: The Yield of Artificial Intelligence (GI Genius) in Lynch Syndrome - A Randomized Tandem-colonoscopy Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-20-6956-IL-CTIL
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-11

CONDITIONS: Lynch Syndrome
Keywords: lynch syndrome; artificial intelligence; tandem colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Artificial Intelligence

STUDY DESIGN:
Intervention Model Description: comparison of 2 groups of patients undergoing tandem colonoscopy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- high-definition white-light endoscopy (No Intervention): patients undergoing first and second colonoscopy with high-definition white-light endoscopy
- artificial intelligence (Active Comparator): patients undergoing first colonoscopy with high-definition white-light endoscopy and second colonoscopy with artificial intelligence
  Interventions: Diagnostic Test: artificial intelligence

INTERVENTIONS:
Diagnostic Test: artificial intelligence — patients will undergo tandem colonoscopy with artificial intelligence
  Arms: artificial intelligence

SUMMARY:
We aim to investigate the incremental detection rate of polyps using AI- assisted colonoscopy compared with high-definition white-light endoscopy (HD-WLE).

We will conduct a single-center randomized tandem colonoscopy trial of patients with Lynch syndrome with and without AI. Patients will undergo tandem colonoscopy, the second colonoscopy with either HD-WLE or an AI- assisted device.

DETAILED DESCRIPTION:
We will include patients with a known pathogenic variant (PV) / likely PV in one of the MMR genes, who are undergoing endoscopic screening and surveillance in our institute. Patients will undergo a first colonoscopy with HD-WLE, and will be randomized at 1:1 ratio to undergo a second colonoscopy with either HD-WLE or an AI- assisted device. All visualized polyps will be removed and size, histology and numbers of polyps detected on each exam will be recorded. We will evaluate the adenoma detection rate and polyp detection rate in each arm and the number of adenomas / polyps in each arm.

ELIGIBILITY:
Inclusion Criteria:

* patients with a known pathogenic variant in one of the mismatch repair genes, who are undergoing endoscopic screening and surveillance in our institute

Exclusion Criteria:

* patients < 18 years old
* lack of informed consent
* concomitant inflammatory bowel disease
* previous total colectomy
* inadequate bowel cleansing (Boston Bowel Preparation Scale (BBPS) ≤5 or < 2 in one of the 3 segments)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-03 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
adenoma incremental detection rate | At the date of enrollment, from the start of colonoscopy until the end of the colonoscopy, in which number of lesions will be detected.
  per lesion analysis, the incremental detection rate will be calculated, defined as the number of lesions detected during the second colonoscopy divided by the total number of lesions detected during first and second colonoscopy combined.

SECONDARY OUTCOMES:
incremental detection rate for advanced neoplasia and any polyp | At the date of enrollment, from the start of colonoscopy until the end of the colonoscopy.
  per lesion analysis, the incremental detection rate for advance neoplasia and any polyp. In the per patient analysis, the increment in adenoma detection rate and any polyp detection rate.
The increment in adenoma detection rate / polyp detection rate | At the date of enrollment, from the start of colonoscopy until the end of the colonoscopy.
  per lesion analysis, the incremental detection rate for advance neoplasia and any polyp. In the per patient analysis, the increment in adenoma detection rate and any polyp detection rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No